CLINICAL TRIAL: NCT05624996
Title: Phase III Prospective Randomized Trial of Primary Lung Tumor Stereotactic Body Radiation Therapy Followed by Concurrent Mediastinal Chemoradiation for Locally-Advanced Non-Small Cell Lung Cancer
Brief Title: Testing the Addition of High Dose, Targeted Radiation to the Usual Treatment for Locally-Advanced Inoperable Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-LU008; NCI-2022-08263 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-LU008 (Other: NRG Oncology); NRG-LU008 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-11-04; First posted 2022-11-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Lung Non-Small Cell Carcinoma; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; durvalumab; Immunoglobulin G; Disulfides; Etoposide; Radiotherapy, Image-Guided; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; osimertinib; Paclitaxel; Pemetrexed; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (image guided RT, chemotherapy, immunotherapy) (Active Comparator): Patients undergo conventional IGRT and receive usual care chemotherapy consisting of paclitaxel IV followed by carboplatin IV Q7D during radiotherapy or pemetrexed IV followed by carboplatin IV every 21 days during radiotherapy or etoposide IV on days 1 to 5 and days 29 to 33 followed by cisplatin IV on days 1, 8, 29, and 36 or pemetrexed IV followed by cisplatin IV every 21 days during radiotherapy. Patients then receive consolidation durvalumab IV every 2 or 4 weeks for up to one year or osimertinib PO QD in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or PET/CT during follow-up.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Etoposide; Radiation: Image Guided Radiation Therapy; Drug: Nab-paclitaxel; Drug: Osimertinib; Drug: Paclitaxel; Drug: Pemetrexed; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Arm II (SBRT, image guided RT, chemotherapy, immunotherapy) (Experimental): Patients undergo SBRT and conventional IGRT and then receive standard-of-care chemotherapy consisting of paclitaxel IV followed by carboplatin IV Q7D during radiotherapy or pemetrexed IV followed by carboplatin IV every 21 days during radiotherapy or etoposide IV on days 1 to 5 and days 29 to 33 followed by cisplatin IV on days 1, 8, 29, and 36 or pemetrexed IV followed by cisplatin IV every 21 days during radiotherapy. Patients then receive consolidation durvalumab IV every 2 or 4 weeks for up to one year or osimertinib PO QD in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or PET/CT during follow-up.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Etoposide; Radiation: Image Guided Radiation Therapy; Drug: Nab-paclitaxel; Drug: Osimertinib; Drug: Paclitaxel; Drug: Pemetrexed; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Radiation: Image Guided Radiation Therapy — Undergo IGRT
  Other Names: IGRT; Image Guided Radiotherapy; image-guided radiation therapy; Image-Guided Radiotherapy
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; ABI007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Naveruclif; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm II (SBRT, image guided RT, chemotherapy, immunotherapy)

SUMMARY:
This phase III trial compares the effect of adding stereotactic body radiation therapy (SBRT) to the usual treatment (conventional image guided radiation therapy [IGRT] and chemotherapy followed by immunotherapy with durvalumab or targeted therapy with osimertinib) versus the usual treatment alone in treating patients with non-small cell lung cancer that has spread to nearby tissue or lymph nodes (locally advanced) and cannot be treated by surgery (inoperable). SBRT uses special equipment to position a patient and deliver radiation therapy to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. IGRT is a type of radiation therapy that creates a picture of the tumor to help guide the radiation beam during therapy, making it more accurate and causing less damage to healthy tissue. Usual chemotherapy used in this trial consists of combinations of the following drugs: cisplatin, carboplatin, paclitaxel, nab-paclitaxel, pemetrexed, and etoposide. Cisplatin and carboplatin are in a class of medications known as platinum-containing compounds. Cisplatin works by killing, stopping, or slowing the growth of tumor cells. Carboplatin works in a way similar to the anticancer drug cisplatin but may be better tolerated than cisplatin. Carboplatin works by killing, stopping, or slowing the growth of tumor cells as well. Paclitaxel is in a class of medications called antimicrotubule agents. It works by stopping the growth and spread of tumor cells. Nab-paclitaxel is an albumin-stabilized nanoparticle formulation of paclitaxel which may have fewer side effects and work better than other forms of paclitaxel. Pemetrexed is in a class of medications called antifolate antineoplastic agents. It works by blocking the action of a certain substance in the body that may help tumor cells multiply. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and deoxyribonucleic acid (DNA) repair and may kill tumor cells. Immunotherapy with durvalumab can induce changes in the body's immune system and can interfere with the ability of tumor cells to grow and spread. Osimertinib is in a class of medications called kinase inhibitors. It works by blocking the action of a protein called EGFR that signals cancer cells to multiply. This helps slow or stop the spread of tumor cells. Adding SBRT to the usual treatment of IGRT with chemotherapy and immunotherapy may be more effective at treating patients with locally-advanced non-small cell lung cancer than giving the usual treatment alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall survival in patients with stage II-IIIC inoperable node-positive non-small cell lung cancer (NSCLC) after image guided, motion-managed conventional radiotherapy to the primary tumor and nodal metastases (Arm 1) or after image guided, motion-managed stereotactic body radiation therapy (SBRT) to the primary tumor followed by conventionally fractionated radiotherapy to nodal metastases (Arm 2) both given with concurrent platinum-based chemotherapy.

II. To compare progression-free survival between the experimental arm (Arm 2) and control arm (Arm 1).

SECONDARY OBJECTIVES:

I. To compare objective response rate (as defined by Response Evaluation Criteria in Solid Tumors [RECIST] version [v] 1.1) between the experimental arm and control arm.

II. To compare the rate of local control between the experimental arm and control arm.

III. To compare patterns of failure (primary, locoregional, or distant) between the experimental arm and control arm.

IV. To compare changes in pulmonary function (forced expiratory volume in 1 second [FEV1] and diffusion capacity of the lung for carbon monoxide [DLCO] assessed at randomization and at 6- and 12- months following completion of radiation therapy) between the experimental arm and control arm.

V. To compare changes in quality of life and patient-reported outcomes assessed from pre-treatment to 3 months following radiation therapy of each treatment arm.

VI. To determine acute and late toxicity profiles of each treatment arm as measured by the Common Terminology Criteria for Adverse Events (CTCAE) v5.

EXPLORATORY OBJECTIVES:

I. To characterize and compare longitudinal quality of life and patient-reported outcomes of each treatment arm.

II. To collect biospecimens at baseline, after SBRT (for Arm 2 patients), during last 2 weeks of chemoradiation, and after first dose of consolidation therapy, to allow for future analyses.

III. To collect 4-dimensional (4D) computed tomography (CT) planning scans and radiation dose to calculate regional lung ventilation and explore pre-treatment 4D-CT based ventilation to predict pulmonary toxicity.

IV. To characterize clinical outcomes, toxicities and changes in pulmonary function and quality of life among patients receiving proton and photon radiotherapy.

V. To develop and characterize a machine learning/artificial intelligence algorithm for radiotherapy planning and/or quality assurance.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo conventional IGRT and receive usual care chemotherapy consisting of paclitaxel intravenously (IV) followed by carboplatin IV weekly (Q7D) during radiotherapy or pemetrexed IV followed by carboplatin IV every 21 days during radiotherapy or etoposide IV on days 1 to 5 and days 29 to 33 followed by cisplatin IV on days 1, 8, 29, and 36 or pemetrexed IV followed by cisplatin IV every 21 days during radiotherapy. Patients then receive consolidation durvalumab IV every 2 or 4 weeks for up to one year or osimertinib orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or positron emission tomography (PET)/CT during follow-up.

ARM II: Patients undergo SBRT and conventional IGRT and then receive standard-of-care chemotherapy consisting of paclitaxel IV followed by carboplatin IV Q7D during radiotherapy or pemetrexed IV followed by carboplatin IV every 21 days during radiotherapy or etoposide IV on days 1 to 5 and days 29 to 33 followed by cisplatin IV on days 1, 8, 29, and 36 or pemetrexed IV followed by cisplatin IV every 21 days during radiotherapy. Patients then receive consolidation durvalumab IV every 2 or 4 weeks for up to one year or osimertinib PO QD in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or PET/CT during follow-up.

Patients are followed up every 3 months for 1 year, every 6 months during years 2 and 3, and then yearly after that for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of non-operable stage IIB or III, node positive (American Joint Committee on Cancer [AJCC] eighth edition) non-small cell lung cancer (NSCLC) with known PD-L1 status prior to registration

  * Patients must have an identified primary tumor and at least one nodal metastasis (peribronchial/hilar/intrapulmonary, mediastinal/subcarinal, supraclavicular/scalene)
  * Up to 4 cycles of systemic therapy received prior to registration for the current study cancer is allowable; any prior chemotherapy for a different cancer is also permissible
  * Patients who refuse surgery, in addition to those who are technically unresectable or medically inoperable, are eligible.
  * Patients with separate tumor nodules in the same lobe of the primary tumor are eligible
* The patient must be deemed clinically appropriate for curative intent definitive combined modality therapy, based on the following staging assessments:

  * History/physical examination prior to registration;
  * Magnetic resonance imaging (MRI) scan of the brain (preferred) or CT scan of the brain (if available, contrast is preferred for all neuroimaging) prior to registration;
  * CT chest with IV contrast (if contrast is available and unless contraindicated, such as for abnormal kidney function) prior to registration. PET/CT may be used if the CT portion is of identical diagnostic quality as achieved in a stand-alone CT
* No evidence of distant metastases based on FDG PET/CT scan obtained within 60 days of registration
* Primary tumor =< 7 cm
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Hematologic function (e.g. platelets, leukocytes, hemoglobin) amenable, at the discretion of the treating physician, to allow for treatment with chemotherapy and concurrent radiation therapy
* Creatinine clearance >= 25 mL/min by the Cockcroft-Gault (C-G) equation
* Subjects with non-malignant pleural effusion are eligible provided the effusion is not known or demonstrated to be an exudative effusion

  * If a pleural effusion is present, the following criteria must be met to exclude malignant involvement:

    * When pleural fluid is visible on both the CT scan and on a chest x-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative;
    * Effusions that are minimal (i.e., not visible on chest x-ray) that are too small to safely tap are eligible
* Medical history consistent with the patient being amenable, at the discretion of the treating physician, to allow for treating with consolidation immunotherapy. Patients with known EGFR/ALK/other driver mutation at the time of registration are eligible, and these patients can be treated with consolidation systemic therapy at the discretion of the treating physician
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Negative pregnancy test =< 14 days prior to registration for participants of childbearing potential
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Prior radiotherapy to the study cancer (local recurrence). Prior radiotherapy for a different cancer/condition to the region of the study cancer that would result in overlap of radiation therapy fields that is determined by the treating physician to impede the treatment of the study malignancy
* Patients without identifiable primary tumor and at least 1 pathologically enlarged lymph node are not eligible (T3-4N0 or T0N1-3 patients are not eligible). At least 1 radiographically-involved lymph node is required, but pathologic confirmation of involvement is not mandated
* Centrally located primary tumor < 2 cm from involved nodal disease that would result in significant overlap of the primary SBRT and nodal radiation fields. This does not include proximity to involved segmental and subsegmental lymph nodes (levels 13 and 14) that would not result in overlap of dose to the proximal bronchial tree or esophagus. Centrally located is defined as within or touching the zone of the proximal bronchial tree, which is a volume 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus right and left lower lobe bronchi)
* Participants who are pregnant or unwilling to discontinue nursing
* Participants of childbearing potential (participants who may become pregnant or who may impregnate a partner) unwilling to use highly effective contraceptives during therapy and for the Food and Drug Administration (FDA)-labeled contraception timeframe required after the final dose of the selected systemic therapy regimen, because the treatment in this study may be significantly teratogenic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2031-10-15 (Estimated); Study Completion 2031-10-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Time between date of randomization and date of death due to any cause, assessed up to 8 years
  Non-inferiority (NI) between arm 2 and arm 1 (reference level) will be evaluated by comparing the upper bound of the 95% confidence interval for the hazard ratio to the pre-specified NI margin. NI of arm 2 will be concluded if the upper bound of the confidence interval is equal to, or falls below, the pre-specified margin at the final analysis. When evaluating the NI of arm 2 in OS, a Cox proportional hazards (PH) model stratified by stratification factors will be used to compute the hazard ratio and associated 95% confidence interval (CI). OS rates will be estimated using the Kaplan-Meier method. If the NI of arm 2 in OS is demonstrated, the superiority of arm 1 in OS will be tested at 1-sided significance level of 0.025 using a stratified log-rank test by adjusting for stratification factors.
Progression-free survival (PFS) | Time between date of randomization and first date of documented progression or death due to any cause, assessed up to 8 years
  The PFS analysis will be conducted using the same methods and stratification factors as the OS analysis. The superiority of arm 2 in PFS will be tested at 1-sided significance level of 0.025 using a stratified log-rank test by adjusting for stratification factors. In the event that the NI of OS is not established, statistical inference of PFS will be considered exploratory in nature only. A Cox PH model stratified by stratification factors will be used to compute the hazard ratio and associated 95% CI.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 8 years
  ORR (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) is defined as the number (%) of patients with at least 1 visit response of complete response (CR) or partial response (PR) and will be based on all randomized patients who have measurable disease. Therefore, data obtained up until progression, or the last evaluable assessment in the absence of progression, will be included in the assessment of ORR. The ORR will be compared between arm 2 versus arm 1 using a Fisher's exact test. A binary response variable for ORR will be used for the analysis with the categories of CR and PR versus stable disease, progressive disease and inevaluable.
Time to progression | Up to 8 years
  Local control also known as time to progression will be defined as freedom from local progression, in which a failure is defined as intrathoracic tumor progression (failure in the lobe of the primary tumor or mediastinal lymph nodes) by RECIST 1.1 criteria. Local control will be analyzed as competing risks data based on cause-specific hazards approaches, where deaths without local failure will be considered as a competing event and analyzed as "censoring" of local failure. The rates at various timepoints (e.g., every 6 months after randomization) and medians of PFS for each arm will be estimated using the Kaplan-Meier method. The associated 95% CI will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Results from an unstratified analysis will also be provided.
Time to primary, locoregional, or distant failure | Up to 8 years
  Competing risks analysis will be used to analyze times to primary failure, locoregional failure and distant failure as the first failure. Competing events include primary failure, locoregional failure, distant failure and deaths without any failures. Rates at various timepoints (i.e., every 6 months after randomization) for each arm will be estimated using the cumulative incidence function. The associated 95% CI will be calculated using the Delta method and based on a log-log transformation applied on the estimated cumulative incidence functions. Statistical inferences of the development of each failure between arms will be based on cause-specific hazards using the log-rank test and Cox proportional hazard model. In addition, Gray's test and the Fine-Gray model will also be used to provide statistical inferences between arms based on cumulative incidence functions and subdistribution hazards.
Changes in pulmonary function | From randomization to 6 months or 12 months
  Includes forced expiratory volume in 1 second (FEV1) and diffusion capacity of the lung for carbon monoxide (DLCO). Changes in pulmonary function (FEV1 and DLCO) will be summarized with descriptive statistics, and compared with Wilcoxon rank-sum test. The descriptive statistics of changes in FEV1 and diffusion capacity before and after treatment will be reported by treatment arm and by response categories (complete response; partial response; stable disease; progressive disease). Linear regression will be used to model changes with adjustment for treatment arms and possibly other baseline covariates, if applicable. The grade 3-5 NRG Oncology Pulmonary Toxicity Scale for changes will be reported with the frequency and grade by arm. Logistic regression will be used to model the distribution of the NRG Oncology Pulmonary Toxicity Scale by arms with and without adjustment for covariates.
Patient reported outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | At 3, 12, and 24 months
  Adverse events will also be assessed using PRO-CTCAE items. The PRO-CTCAE is a patient-reported outcome measurement system developed to characterize the frequency, severity, and interference of symptomatic treatment toxicities. Items are scored on a Likert scale. For each symptom and each domain (i.e., frequency, severity, and interference), counts and frequencies will be summarized for the worst score experienced by the patient by the treatment arm. In addition, a composite grading algorithm (Basch 2021) will be used to derive a single numerical grade for each adverse event scored using PRO-CTCAE. PRO-CTCAE, the frequency of acute grade >= 3 patient-reported toxicity will be compared to the corresponding rate of clinician-scored toxicity using a chi-square test or Fisher exact test, as appropriate. Distributions of clinician-reported and patient-reported adverse events will also be compared across study arms.
Functional Assessment of Cancer Therapy Lung (FACT-L) and Trial Outcome Index (TOI) | At 3, 12, and 24 months
  FACT-L and TOI is a measure that sums the functional well-being (FWB - 7 items), physical well-being (PWB - 7), and the lung cancer subscale (LCS - 9 items) of FACT-L. Questionnaire trial outcome index deterioration rates at 3 months and associated 95% confidence interval will be calculated for each treatment group, based on all randomized subjects. In addition, to explore if higher QOL scores will be maintained at 12 and 24 months from the end of radiotherapy as well, longitudinal data analysis will also be performed to characterize the trend of scores over time across the two treatment groups using hierarchical formulation of the linear mixed model. The Clopper-Pearson method will be used for calculating 95% CI. The deterioration rates of each arm will also be compared using Cochran-Mantel-Haenszel Test, stratified by PD-L1 expression and T-stage.
European Quality of Life Five Dimension (EQ-5D) scale | At 3, 12, and 24 months
  Subjects' overall health state on a visual analog scale (EQ-VAS) at each assessment time point will be summarized using descriptive statistics by treatment group, as randomized. Proportion of subjects reporting problems for the five EQ-5D dimensions at each assessment time point will be summarized by level of problem and by treatment group, as randomized. Percentages will be based on number subjects assessed at assessment time point.
Incidence of adverse events | Up to 8 years
  For each patient, the maximum severity reported will be used in the summaries. Adverse events will be summarized regardless of relationship to protocol treatment as assessed by the investigator. Treatment-related adverse events using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) will be presented in statistical analysis reports/publications in CTCAE version 5. Adverse event rates will be reported with the frequency and severity (e.g., type, grade, and attribution) by arm.

OTHER OUTCOMES:
Clinical outcomes | Up to 8 years
  Descriptive analyses will be reported, based on corresponding analysis plans within patients who actually receive proton and photon radiotherapy (e.g., per-protocol population), respectively.
Functional mean lung dose | Up to 8 years
  Collection of 4-dimensional (4D) computed tomography (CT) planning CTs and calculation of radiation dose to regional lung ventilation will be performed among randomized patients with 4D CT planning CTs. To evaluate functional dose metrics, ventilation maps will be registered to the average 4DCT reference frame. Functional dose metrics and standard dose metrics will be calculated and evaluated. Functional mean lung dose will be defined as the mean dose delivered to functional lung. Dose to total lung and dose to functional lung will then be correlated with pulmonary toxicity including grade 2 or higher radiation pneumonitis or any grade 3 or higher cough, dyspnea, hypoxia or respiratory failure. Logistic regression models will be used to explore the correlation between pulmonary toxicity and functional mean lung dose.
Incidence of toxicities | Up to 8 years
  Descriptive analyses will be reported, based on corresponding analysis plans within patients who actually receive proton and photon radiotherapy (e.g., per-protocol population), respectively.
Changes in pulmonary function | Up to 8 years
  Descriptive analyses will be reported, based on corresponding analysis plans within patients who actually receive proton and photon radiotherapy (e.g., per-protocol population), respectively.
Changes in quality of life | Up to 8 years
  Descriptive analyses will be reported, based on corresponding analysis plans within patients who actually receive proton and photon radiotherapy (e.g., per-protocol population), respectively.
Development and characterization of a machine learning/artificial intelligence (AI) algorithm for radiotherapy planning and/or quality assurance | Up to 8 years
  Assessment will focus on four key areas: tumor volume contouring score, organs-at-risk contouring score, tumor volume dose-volume analysis score, and organs-at-risk dose-volume analysis score. Each area will be scored as per protocol: acceptable variation, unacceptable variation, or not evaluable. Cases deemed not evaluable will be considered as such, regardless of the reviewer. The scores generated by the AI algorithm will be compared with those from radiation oncologists, ensuring the AI algorithm adheres to the contours. The sensitivity of the AI algorithm, indicating its ability to detect deviations from the protocol, will be calculated. The AI algorithm will be refined until its sensitivity exceeds 95%. Inter-rater reliability between the AI algorithm and the radiation oncologists will be assessed using Cohen's κ. Concordance and discordance frequencies will also be recorded.
Treatment effect and confidence intervals by sex | Up to 8 years
Treatment effect and confidence intervals by race | Up to 8 years
Treatment effect and confidence intervals by ethnicity | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Simone, Principal Investigator — NRG Oncology
Locations (466):
- United States (465):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Gulf Health Hospitals Inc/Infirmary Cancer Care - Malbis, Daphne, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Gulf Health Hospitals Inc/Infirmary Cancer Care - Saraland, Saraland, Alabama
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Hamilton Medical Center - Peeples Cancer Institute, Dalton, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Alton Memorial Hospital, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Wilmot Cancer Center at Batavia, Batavia, New York
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - New York Proton Center, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Westchester Medical Center, Valhalla, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Levine Cancer Institute - Rutherford, Forest City, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Novant Health Breast Surgery - Greensboro, Greensboro, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Levine Cancer Institute - Union West, Matthews, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Wake Forest Baptist Health - Hematology Oncology - Statesville, Statesville, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Lancaster Radiation Therapy Center, Lancaster, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Virginia Mason Medical Center, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Heinzerling JH, Mileham KF, Robinson MM, Symanowski JT, Induru RR, Brouse GM, Corso CD, Prabhu RS, Haggstrom DE, Moeller BJ, Bobo WE, Fasola CE, Thakkar VV, Pal SE, Gregory JM, Norek SL, Begic XJ, Kesarwala AH, Burri SH, Simone CB 2nd. Primary lung tumour stereotactic body radiotherapy followed by concurrent mediastinal chemoradiotherapy and adjuvant immunotherapy for locally advanced non-small-cell lung cancer: a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2025 Jan;26(1):85-97. doi: 10.1016/S1470-2045(24)00573-4. Epub 2024 Nov 29. PMID 39615497